CLINICAL TRIAL: NCT07097766
Title: The Effect of Health Belief Model-Based Education and Motivational Interviewing on Human Papillomavirus (HPV) Infection Knowledge Level and HPV Vaccine Awareness Among Women
Brief Title: The Effect of Health Belief Model-Based Education and Motivational Interviewing on HPV (Human Papilloma Virus) Knowledge and Vaccine Awareness in Women
Acronym: HPV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Seda Ayyıldız, Seda Ayyıldız (Doctoral Student), Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: SAYYILDIZ2025HPV
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Human Papillomavirus Infection
Keywords: HPV; Human Papillomavirus; HPV Vaccine; Health Belief Model; Motivational Interviewing; Vaccine Awareness; Women's Health; Cervical Cancer Prevention
MeSH Terms: conditions — Papillomavirus Infections | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either an intervention group receiving HBM-based education and motivational interviewing, or a control group receiving no intervention. Outcomes will be assessed before and after the intervention.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcomes assessors were blinded to group assignments. However, the intervention provider was aware of group allocation due to the nature of the educational intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Behavioral: "HBM-Based Education and Motivational Interviewing"
- Control Group (No Intervention): This group will not receive any educational intervention or motivational interviewing. Standard care or routine health information will be provided as per usual practice.

INTERVENTIONS:
Behavioral: "HBM-Based Education and Motivational Interviewing" — This intervention consists of a structured 3-session educational program and motivational interviews based on the Health Belief Model (HBM). It aims to increase knowledge about HPV infection and improve HPV vaccination awareness among women aged 18-45.
  Arms: Intervention Group

SUMMARY:
This study aims to evaluate the effect of an educational intervention based on the Health Belief Model (HBM) combined with motivational interviewing on women's knowledge about Human Papillomavirus (HPV) infection and their awareness of HPV vaccination. The study will be conducted among women aged 18-45 who have not received the HPV vaccine. Participants in the intervention group will receive structured education and motivational interviews, while the control group will receive no intervention. Changes in HPV knowledge and vaccine awareness will be measured before and after the intervention using validated scales. The goal is to improve preventive behaviors and increase vaccine uptake through behavior-based education.

DETAILED DESCRIPTION:
This randomized controlled trial is designed to assess the impact of education and motivational interviewing grounded in the Health Belief Model (HBM) on women's knowledge regarding HPV and awareness of the HPV vaccine. The study population consists of 18-45-year-old literate women who have not previously received HPV vaccination.

Participants will be randomly assigned to either an intervention group or a control group. The intervention group will receive a 3-session structured education program based on HBM constructs (perceived susceptibility, perceived severity, perceived benefits, perceived barriers, cues to action, and self-efficacy), supported by motivational interviewing techniques. The control group will receive no intervention.

Data collection will include pre- and post-intervention assessments using a validated HPV knowledge scale and vaccine awareness questionnaire. The expected outcome is a statistically significant improvement in knowledge and awareness in the intervention group.

This study aims to contribute to public health efforts in HPV prevention and vaccination promotion by utilizing a behavioral model in community education.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 18-45 years

Voluntary participation and providing informed consent

Not previously vaccinated against HPV

Ability to attend all three educational and motivational interview sessions

Literacy sufficient to complete study questionnaires

Exclusion Criteria:

* Women under 18 or over 45 years old

Prior HPV vaccination

Cognitive or psychiatric conditions that hinder participation

Currently participating in another HPV-related education or intervention study

Inability to attend all sessions of the intervention program

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — only individuals who identify as female and meet the age criteria will be eligible to participate in the study
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
HPV Knowledge Score | 4 weeks after the intervention
  Participants' total score on an HPV knowledge questionnaire designed to assess understanding of HPV infection, transmission, and prevention.

SECONDARY OUTCOMES:
HPV Vaccination Awareness Score | 4 weeks after the intervention
  Participants' awareness level regarding HPV vaccination, measured using a structured 10-item survey.

CONTACTS AND LOCATIONS:
Locations (1):
- Zeynep Kamil Kadın ve Çocuk Hastalıkları Eğitim ve Araştırma Hastanesi, Üsküdar, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
IPD and supporting documents will be available starting 6 months after the publication of the primary study results and will remain available for 5 years.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD and supporting documents will be available starting 6 months after the publication of the study results and will remain available for 5 years.
Access Criteria: Qualified researchers may request access to the individual participant data by contacting the principal investigator. Access will be granted upon reasonable request and approval of a data sharing agreement.